CLINICAL TRIAL: NCT01108120
Title: The Therapeutical Role of Continuous Intra-femoral Artery Infusion of Urokinase on Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: q9jhrvf3-2
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot ulcer; artery mini-pump; continuous infusion of urokinase; femoral artery
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous intra-femoral thrombolysis group (Experimental): Continuous intra-femoral injection urokinase was taken by a mini-pump in 100 diabetic foot ulcers (Wegnar 2 ~ 4 stage) for 7 - 9 days.Then they receive conventional therapy. The healing rate of foot ulcers is observed during hospitalization period. At 1, 4 and 8 year during follow up, the recurrence rate of diabetic foot ulcers are observed.
  Interventions: Drug: continuous intra-femoral thrombolysis group
- conventional therapy group (Active Comparator): Conventional therapy group receives an intravenous injection of prostaglandin E1 20 ug per day. The follow up was taken for 8 years.
  Interventions: Drug: Conventional therapy group

INTERVENTIONS:
Drug: continuous intra-femoral thrombolysis group — Firstly, 20 0000 u urokinase is injected to the diseased foot via catheter. Then, continuous injection of urokinase via femoral artery by a artery mini-pump (100 ml 0.9% sodium chloride + 100 0000 unit urokinase at a rate of 4 ml per hour) is taken for 7 - 9 days.
  Arms: continuous intra-femoral thrombolysis group
Drug: Conventional therapy group — All patients receive an intravenous injection of prostaglandin E1 20 ug per day during hospitalization period.
  Arms: conventional therapy group

SUMMARY:
* Diabetic foot ulcers (DFU) are one of the chronic consequences of diabetes which constitute the most important cause of non-traumatic amputation of the inferior limbs. Patients with diabetes are 22 times more likely to have foot ulceration or gangrene than nondiabetics，while foot ulceration precedes 85% of lower-extremity amputation.
* Three factors combine to promote tissue necrosis in diabetic feet: ischemia, neuropathy and trauma. Among them, ischemia peripheral arterial disease may play the important roles in the development of DFU. Moreover, diffuse vascular disease is the main characteristics, and thus it becomes difficult for treatment by using arterial bypass or balloon angioplasty. Therefore, we hypothesized that continuous arterial thrombolysis may be an effective therapy in diabetic foot. The purpose of this study is to investigate the effectiveness and safety of continuous intra-femoral artery injection of urokinase by micro-artery-pump in diabetic ulcers.

DETAILED DESCRIPTION:
* We select 200 diabetic patients with Wagner grade 1 ~ 3 foot ulcers. They are divided into two groups randomly: thrombolysis group and control group, 100 cases in each group.
* After diabetic dietary advice, all patients receive insulin therapy to control blood glucose within a range of 5 - 10 mmol/L. Then the patients receive conventional care for their ulcers. To remove extensive callus and necrotic tissue, wound debridement was performed. Broad spectrum antibiotics are prescribed if ulcers show clinical signs of infection. Adjustments to the treatment are performed when indicated on the basis of microbiologic cultures and sensitivity testing.
* The conventional group patients receive an intravenous injection of prostaglandin E1 (20 ug per day)until the healing of ulcers or discharged from hospital. In the continuous intra-femoral thrombolysis group, first of all, a ultrasound Doppler examination of vessels including artery and venous of lower limbs were performed. To avoid pulmonary infarction, a filtrator is placed in the inferior vena cava before the thrombolysis process if ultrasound results show venous thrombosis. Then insert a percutaneous artery canal from femoral artery in another lower limb into the distal of popliteal artery as far as possible. After finishing this process, the outside part of this artery canal is fixed at thigh, and the patients must keep in supine position in the bed.Firstly,20 0000 ~ 40 0000 units urokinase is injected via the catheter to diseased foot. Then, continuous infusion urokinase via femoral artery by an artery pump (100 ml 0.9% sodium chloride + 100 0000 unit urokinase at a rate of 4 ml per one hour) for 7 - 10 days. Finally, patients receive an intravenous injection of prostaglandin E1 (20 ug per day)until the healing of ulcers or discharged from hospital.
* The healing rate of foot ulcers, the time of ulcers, neuropathy symptoms, the period of hospitalization are compared between the two groups during hospitalization.
* The recurrence rate of foot ulcers, cardiovascular events, death from all causes are compared between two groups at 1, 4, 8 years during follow up.

ELIGIBILITY:
Inclusion Criteria:

* diabetic foot ulcer
* < = 80 years old
* diabetic foot ulcer wegnar 2-4 stage

Exclusion Criteria:

* Wagner grade 0,1 and grade 5
* severe coronary, cerebral, renal vascular as well as severe liver diseases, malignant neoplasms
* bleeding individuals
* > 80 years old
* heart failure (NYHA 3,4)
* cancer

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-05; Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
healing rate of diabetic foot ulcers | < half a year
  During hospitalization, the healing rate of foot ulcers is observed.
The recurrence rate of diabetic foot ulcers | 8 years
  During the 8 years of follow up period, recurrence rate of diabetic foot ulcers are observed at 1, 4, 8 year.

SECONDARY OUTCOMES:
cardiovascular events during the follow up period | 8 years
  During the follow up period of 8 years, the cardiovascular events, death from all causes are observed at 1, 4 and 8 year.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of Central theater Command, Wuhan, Hubei, China

REFERENCES:
- [Derived] Tong J, Zhang J, Xiang L, Li S, Xu J, Zhu G, Dong J, Cheng Y, Ren H, Liu M, Yue L, Xiang G. Continuous intrafemoral artery infusion of urokinase improves diabetic foot ulcers healing and decreases cardiovascular events in a long-term follow-up study. BMJ Open Diabetes Res Care. 2024 Jan 12;12(1):e003414. doi: 10.1136/bmjdrc-2023-003414. PMID 38216296